CLINICAL TRIAL: NCT01617512
Title: Study Accelerometer Signals to Measure Daily Activities: a Pilot Study
Brief Title: Study Accelerometer Signals to Measure Daily Activities (SASMDA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdministrateurCIC (Other)
Collaborators: TIMC-IMAG (Other); Laboratory TIMA (Unknown); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor-Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DCIC 1116
Record Dates: First submitted 2011-12-15; First posted 2012-06-12 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Urinary Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: LIS302DL accelerometer — Recording for 24 hours accelerations related to daily physical activity of the patient.

SUMMARY:
The purpose of this study is to determine if it is possible to identify activities in the daily accelerometer measures of a person with urinary disorders.

ELIGIBILITY:
Inclusion Criteria:

* man
* patients fitted with artificial urinary sphincter
* patients affiliated to social security or similar regime

Exclusion Criteria:

* patient do not speak french
* patient unable to express his consent
* patient hospitalize without consent
* patient under legal protection
* patient deprived of liberty

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with urinary disorders for which it is possible to identify automatically activities among all the daily accelerometer data. | 6 months
  Intrinsic characteristics (sensitivity, specificity, ROC curve) of the test for detecting in automated way the activities among all the daily accelerometer data

SECONDARY OUTCOMES:
Score of satisfaction with the use of the medical device, assessed by the patients | 6 months
  Score between 0 and 10, takes into account the feasibility of the proposed approach and the patient felt the importance of this feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Moreau-gaudry, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France